CLINICAL TRIAL: NCT07184541
Title: The Effect of a Nurse-led Daily Weight Monitoring Intervention (Wake and Weigh) on Heart Failure Quality of Life and Self-care
Brief Title: A Nurse-Led Weight Monitoring Intervention For Heart Failure Quality of LIfe and Self-Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lee Anne Siegmund (Other)
Responsible Party: Sponsor-Investigator, Lee Anne Siegmund, Senior Nurse Scientist, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-976
Record Dates: First submitted 2025-02-23; First posted 2025-09-22 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure
Keywords: Heart Failure; Self-care; Quality of life; Weight
MeSH Terms: conditions — Heart Failure; Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wake and Weigh Intervention (Active Comparator): The Wake and Weigh weight log in addition to usual care
  Interventions: Behavioral: Wake and Weigh
- Control (Active Comparator): The heart failure handbook (routinely given for first heart failure admission), and heart failure education per usual care
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Wake and Weigh — The Wake and Weigh tool includes the patient's dry weight and instructions for daily weight monitoring. Participants in the intervention group will be instructed on the use of the tool. While in the hospital, weight is being managed by the healthcare team, so the goal during hospitalization is to educate the patient on what to do once discharged, and to recognize changes in weight.
  Arms: Wake and Weigh Intervention
Behavioral: Usual care — The usual care group will receive the heart failure handbook that is routinely given to heart failure patients.
  Arms: Control

SUMMARY:
Ongoing self-care for heart failure is essential to avoid complications and hospitalization. Supportive strategies are needed; however, patients with heart failure may find many interventions complicated and overwhelming. The purpose of this pilot study is to implement a simple weight tracking tool (Wake and Weigh) to affect self-care and quality of life in a population of older adults with heart failure. This will be a randomized controlled pilot trial to test the methods to be used in a larger randomized controlled trial. The Self-care in Heart Failure Index and Kansas City Cardiomyopathy Questionnaire surveys will be given at admission and four weeks after discharge. The Wake and Weigh tool is designed to help patients track weight in the hospital and following discharge. Feasibility endpoints will be summarized descriptively.

DETAILED DESCRIPTION:
Research question: Are the methods used in a pilot study that is designed to implement a nurse-led daily weight monitoring intervention, appropriate for a larger study to be conducted later, which will test the intervention's effect on self-care and quality of life among older adults with heart failure, compared to those who receive routine care? It may be unrealistic to expect patients to have the agency to perform adequate self-care when they are living with activity-limiting symptoms, and perceive that heart failure (HF) self-care instructions are complicated. Given that HF symptoms interfere with the ability to perform self-care, it is vital to concurrently address symptoms and self-care, while also attempting to reduce information overload. Therefore, the purpose of this pilot study is to implement a simple weight tracking tool to affect HF self-care and HF quality of life (using a measure that focuses on symptoms and quality of life) in a population of adults age 55 years and older who have HF, and test the methods to be used in a larger study.

1. The primary (exploratory) aims of this pilot study are to test methods to be used in a future randomized controlled trial:

   1. Determine intervention fidelity by 1) examining unintended variations in intervention implementation by nurse investigators, and 2) evaluating use (versus no use) of the Wake and Weigh tool by participants.
   2. Determine the feasibility of recruitment by assessing how long it takes to recruit 10% of the anticipated larger study sample size.
   3. Determine the feasibility of randomization and retention for each group.
   4. Test the use and appropriateness of the SCHFI and KCCQ in a population of recently discharged adults aged 55 years and older who have HF who had been admitted to a small regional hospital.

   a. Test the appropriateness of the chosen measures by i. Determining percentage of completed SCHFI and KCCQ
2. The secondary aim for this study is to test participants' HF self-care and quality of life i. Reporting test scores for the SCHFI and KCCQ (descriptive) ii. Reporting results of additional questions on confidence, belief, and likelihood of use for Wake and Weigh tool (see variable list) iii. Reporting change in test scores if sample size allows. The setting for this study is a 126-bed regional hospital (Cleveland Clinic, Avon Hospital) in Northeast, Ohio. The hospital inpatient areas include adult medical-surgical units and a 12-bed medical intensive care unit. All inpatient areas in the hospital care for patients with HF. Participants for this study will be selected from a population of adult inpatients at the study site who have a new or existing diagnosis of HF.

The intervention for this study will be the introduction and implementation of the Wake and Weigh tool, which will be provided on hospital admission to patients with HF who are randomized to the intervention group. Currently, usual care education for weight and fluid management is delivered utilizing a HF handbook. Although the handbook is available, patient use of the weight record in the handbook is inconsistent. The handbook is given only on initial HF admission, whereas the Wake and Weigh tool is designed as an additional visual management tool, to remind patients to weigh upon waking and to monitor for weight changes. It is designed for any and all admissions for patients with HF. Further, the Wake and Weigh tool is designed to help patients learn to recognize weight changes through daily weighing, using nurse-led role modeling while they are hospitalized and for easy use at home after discharge.

The nurse investigators will introduce the Wake and Weigh tool to admitted patients and will educate them on the importance of weighing daily (See Wake and Weight script). They will be encouraged to use it daily while in the hospital, and at home after discharge. Because it is a short, paper tool, it can be easily taken to provider follow-up appointments. The Wake and Weigh tool includes the patient's dry weight and instructions for daily weight monitoring. Patients and/or family members can log the date, time, and weight value beginning in the hospital and maintain the same routine after discharge. It will also include the cardiologist or PCP contact information depending on which provider is managing the patient's HF and follow up care upon discharge. Participants in the intervention group will be instructed to 1) use the same scale each day and record their weight on the form, 2) weigh themselves first thing each morning after using the bathroom, and before eating breakfast, and 3) report to their provider if there is an increase or decrease in four pounds or more when compared to dry weight (discharge weight). While in the hospital, weight is being managed by the healthcare team, so the goal during hospitalization is to educate the patient on what to do once discharged, and to recognize changes in weight.

Pilot feasibility

1. Intervention fidelity will be determined by 1) nurse investigators' consistent patient education of the Wake and Weigh intervention, and 2) the participant use of the tool.

   First, fidelity will be determined by the number of times it takes for all nurse investigators (n=5) to provide the Wake and Weigh intervention education consistently through role-playing prior to recruiting participants. An intervention checklist will be used and all areas must be complete to be counted. If this can be accomplished in 5 or fewer attempts, the fidelity of the intervention will be considered feasible.

   Post-intervention, the investigators will determine whether the participant used the Wake and Weigh form or not. They will also be asked whether they went to their follow-up visit, whether they took it to their provider and whether they were hospitalized since starting the study; however, this will not be included as an intervention outcome. During the post-intervention phone call, the nurse investigator will ask the participant about Wake and Weigh use (see follow-up calls document). Greater than 70% of participants using the Wake and Weigh form (determined by self-report of weighing and recording weight at least half the time since hospital discharge) will be required to determine that the intervention is feasible for the larger study.
2. Recruitment feasibility will be determined by the length of time (weeks, months) it takes to recruit a minimum sample size (n=42), which 9% of the minimum for a larger study.
3. Randomization and retention feasibility will be determined by the percentage of participants who stay in the assigned group and in the study until completion of exit surveys. Study dropouts will be reported by group. If 70% or more of the control group and 70% or more of the intervention group remain in the study for two weeks or until study follow-up call, randomization will be considered feasible. If 70% or more of all participants remain in the study for two weeks or until study follow-up call, retention will be considered feasible.
4. The appropriateness of the instruments and instrument scores will be determined with internal consistency, percentage of completed surveys (80% of participants complete both surveys=appropriate for a larger study), and survey inter-correlations (surveys correlated at < 0.3). Test scores will be reported descriptively and change in test scores will be reported if minimum sample size or greater is obtained.

Measures

1. Self-care in Heart Failure Index (SCHFI). The SCHFI v7.2-C will be used to measure HF self-care behaviors. It includes 3 scales: Self-Care Maintenance (5-point Likert scale from 1 to 5), Symptom Perception (first 9 items were rated on a 5-point Likert scale, and the last 2 items were responded to as "have not had symptoms," 0 (I did not recognize the symptoms), 1 (not quickly) to 5 (very quickly), and Self-Care Management (5-point Likert scale from 1 to 5 for the first 7 items and a 6-point rating scale for the last item). Symptom perception was found to include monitoring ("listening" to their bodies) and recognition (engage in active behaviors based on interpretation of symptoms) of HF symptoms. Cronbach's alpha for all scales was ≥ 0.70. Participants who were healthier had higher self-care maintenance score (r = -0.19, P = .08) and higher symptom perception scores (r = -0.31, P = .003). A standardized score from 0 to 100 was calculated for each scale, with higher scores indicating better self-care behavior.
2. KCCQ-12. Heart failure quality of life will be measured by the KCCQ-12. The KCCQ-12, a shortened and more feasible version of the KCCQ-23, is a HF specific health related quality of life questionnaire that describes physical limitations and symptoms, quality of life, social interference, and self-efficacy. This 12-item questionnaire uses a Likert scale from 1-5 (1 = every morning, all of the time, every night, or it has extremely limited my enjoyment of life, 5 = never over the past 2 weeks, it has not limited my enjoyment of life at all), and 2 items on a 1-6 scale (1 = extremely limited/severely limited, 6 = limited for other reasons or did not do the activity/does not apply or did not do for other reasons). Higher scores indicate the following: fewer physical limitations, fewer symptoms, better social functioning, and better sense of self-efficacy and higher quality of life, referred to here as HF quality of life. The KCCQ-12 has high correlations with the original scale (>0.93) and high test-retest reliability (>0.76). 16 Items are scored from 0 to 100 with 0 representing the worst and 100 the best possible functional status.
3. Charlson Comorbidity Index. The Charlson Comorbidity Index (CCI) measures the burden of chronic conditions by applying a weight to a list of specific diseases. The original CCI was reduced to 12 diseases, each of which is specified by using ICD-10 codes. The C-statistic for the Quan 12-item CCI was 0.825, indicating very good discrimination for in-hospital mortality prediction. Stepwise increases in the CCI score were associated with increases in mortality for a wide variety of conditions and in multiple versions (p<0.001) of the CCI.

Middle Range Theory. The Wake and Weigh tool is a simple weight monitoring intervention, derived from aspects of Riegel's middle range theory of self-care in chronic illness, including that self-care is a learned process, effective management requires ongoing monitoring, patients need to identify changes in order to act on them appropriately, and maintenance leads to illness stability and optimal quality of life. Consistent with the theory of self-care, the Wake and Weigh tool is designed to help patients 1) learn from nurses' role modeling of the importance of self-care behaviors related to fluid retention (learn), 2) track weight in the hospital and following discharge, (track), 3) recognize changes in weight before complications arise (identify), and 4) establish a sustainable routine for daily weight monitoring (maintain).

Data Collection The unit RNs will be introduced to the study during huddles and a study sign will be hung in break rooms. Only the research team will introduce the Wake and Weigh form using a script and do education surrounding the form (beyond usual care). Patients will be recruited by the study team members. After determining patients with HF have been admitted to the hospital (HF dashboard will be accessed by one of the team members [BM]), potential participants' names and MRNs who fit inclusion, will be added to a password protected EXCEL spreadsheet, accessible only to the research team. A subject ID will be given for each participant in REDCap, a secure data management system, and data will be recorded and stored in REDCap until analysis. The subject ID will be added to paper surveys (SCHFI and KCCQ) until the data has been entered into REDCap. Since admission for those diagnosed while in the hospital will precede HF diagnosis, the time of diagnosis will be used to determine hospital admission. Within 24 hours of admission, a team member will approach potential participants in the privacy of their patient room, explain the study, and obtain signed informed consent. This will then be documented in the data collection form. After consent, participant will be randomized to group (REDCap), and for those in the intervention group, the Wake and Weigh form will be introduced.

The SCHFI and KCCQ paper surveys will be given immediately before randomization (in person). If the patient verbalizes they are too tired to take the surveys, nurse investigator will approach the potential participant up to 2 additional times (no closer than 24 hours between each time to be sensitive to patient fatigue) until patient feels well enough to take the surveys or declines to participate. The participant will be asked to continue to use Wake and Weigh form as instructed throughout admission, and a nurse investigator will check in daily to reinforce the intervention briefly (ask if they are using it and if they have any questions).

Follow-up (post-intervention) will occur 2 weeks (intervention group only) and 4 weeks after discharge (both groups) via phone. For the 2-week follow-up calls, the nurse investigator will ask the intervention group participants if they have any questions about the Wake and Weigh tool.

For the 4-week follow-up call:

1. Did you attend a provider follow-up visit after discharge? yes/no; 1a. If "yes", which provider (specialty)? 2. Did you take your Wake and Weigh form with you to the follow-up visit (intervention group only)? yes/no); 3. Are you confident that you can recognize weight changes before symptoms appear? Yes/no; 4. Did you experience weight changes of 4 pounds or more since beginning this study and if so, when? Yes/no/don't know; Comments ______5. If yes, did you report the weight change to your provider? Yes/no; 5a. If "yes", which provider (specialty)? 6. Do you believe daily weighing is important for preventing hospitalization? Yes/no; 7. Have you had a hospitalization since beginning this study? Yes/no; 8. If "yes", were you admitted to a Cleveland Clinic hospital? Yes/no; 9. Are you likely to continue to use the Wake and Weigh tool on a regular basis? Yes/no (intervention group only). 10. Reason for continuing/not continuing to use Wake and Weigh (intervention group only).

**per patient report

If at any point during contact (in person or on the phone) participant complains to nurse investigator of new or worsening symptoms, the clinical nurse caring for the patient will be notified (while in hospital), and after discharge participant will be referred to provider.

Analysis Plan Primary analysis will be performed using the intent-to-treat population. Patient characteristics will be summarized by group using frequencies and percentages for categorical factors, and means and standard deviations for continuous measures, if normally distributed, and medians and quartiles, otherwise. Feasibility endpoints will be summarized descriptively as the frequencies with percentages or summaries of time measures, as appropriate. Groups will be compared on overall self-care (SCHFI) and quality of life (KCCQ) using analysis of covariance models that adjust for the baseline levels of each outcome measure. Mean differences in outcomes will be estimated and both 95% two-sided confidence intervals and one-sided 90% confidence intervals will be generated to evaluate plausible differences and the feasibility of an 8-point difference based on this study. To evaluate the association between SCHFI and KCCQ, Pearson correlations between tools will be estimated. McDonald's omega will be used to assess internal consistency of each tool. Secondary analyses may include adjustment for patient characteristics that show standardized differences between randomized groups in excess of 0.2. Additionally, if there are issues with adherence to the intervention, similar analyses among those who adhere to the intervention will also be performed. Analyses will be performed using SAS software (version 9.4) or R software (version 4.2). An overall significance level of 0.05 will be assumed for all tests.

Feasibility This pilot study is feasible as designed due to a large number of weekly HF admissions. Also, the research team consists of research-active nurses and members of the research council, and are being mentored by a nurse scientist from nursing research and innovation. This study has received the approval of the hospital's Chief Nursing Officer (CNO) and a letter of support(CNO Avon letter of support document) will be uploaded into Webkit. Additionally, the hospital's CNO has agreed to provide funds for the cost of the KCCQ.

Limitations and Anticipated Problems The main limitation of this pilot study is the possible inability to infer differences between groups. Analysis of group differences is not a primary aim and will only be conducted if greater than minimum sample size is met for both groups. Anticipated problems for this study include difficulties with recruitment and retention. As this is a common problem with randomized controlled trials, a pilot study will be conducted first to determine challenges and make changes in methods to prepare for a larger study.

Protection of Human Subjects This pilot study will be approved by the institutional review board prior to implementation. Further, informed written consent will be obtained from participants in both groups, and they will be assured that they can stop participation in the study at any time. Names and MRNs will be removed and replaced with a subject number prior to analysis. Any collected data on paper, including consents, will be kept in a locked office chosen by the PI, at Avon Hospital's campus, in a locked filing cabinet. All electronic data (REDCap) will be stored on the PI's computer which requires password entry and will be in a folder accessible only to the PI and the research team. Data will be stored for a period of six years after completion of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (55 years or older)
2. New or existing diagnosis of HF (regardless of type or length of time since diagnosis).
3. Being treated for HF signs and/or symptoms during the current hospitalization (any of the following: IV diuretic, fluid restriction, low sodium diet).
4. Must be able to read and communicate in English.
5. Must be able to stand and weigh independently.
6. Must have a scale at home, or ability to obtain one for the study.

Exclusion Criteria:

1. Documented diagnosis of cognitive impairment.
2. A Charlson Comorbidity Index (CCI) of >4. This was chosen to exclude patients more likely to have hospital stays longer than a week. A CCI of >3 was based on research showing a relationship to mortality (Imam et al., 2020), a CCI of ≥ 6 with a 2.8-times higher mortality (Yilmaz & Omurlu, 2019), and likelihood of longer hospital length of stay for patients with HF if CCI >2 (Foraker et al., 2014).

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Project Feasibility-fidelity | From enrollment to the end of treatment at 4 weeks post-discharge
  Determine intervention fidelity by examining unintended variations in intervention implementation by nurse investigators
Project feasibility-use of tool | From enrollment to the end of treatment at 4 weeks post-discharge
  Evaluate use (versus no use) of the Wake and Weigh tool by participants.
Project feasibility-recruitment | From enrollment to the end of treatment at 4 weeks post-discharge
  Assess how long it takes to recruit 10% of the anticipated larger sample size
Project feasibility-randomization | From enrollment to the end of treatment at 4 weeks post-discharge
  Assess retention in each randomized group
Project feasibility-appropriateness of SCHFI | From enrollment to the end of treatment at 4 weeks post-discharge
  Determine percentage of completed SCHFIs
Project feasibility-appropriateness of KCCQ | From enrollment to the end of treatment at 4 weeks post-discharge
  Determine percentage of completed KCCQs

SECONDARY OUTCOMES:
Heart Failure Quality of Life | From enrollment to the end of treatment at 4 weeks post-discharge
  Heart failure quality of life will be collected using Kansas City Cardiomyopathy Questionnaire-12. This 12-item questionnaire uses a Likert scale from 1-5 (1 = every morning, all of the time, every night, or it has extremely limited my enjoyment of life, 5 = never over the past 2 weeks, it has not limited my enjoyment of life at all), and 2 items on a 1-6 scale (1 = extremely limited/severely limited, 6 = limited for other reasons or did not do the activity/does not apply or did not do for other reasons). Higher scores indicate the following: fewer physical limitations, fewer symptoms, better social functioning, and better sense of self-efficacy and higher quality of life, referred to here as heart failure quality of life.
Heart Failure Self-care | From enrollment to the end of treatment at 4 weeks post-discharge
  Change in heart failure self-care test scores will be collected using the Self-care in Heart Failure Index. It includes 3 scales: Self-Care Maintenance (5-point Likert scale from 1 to 5), Symptom Perception (first 9 items were rated on a 5-point Likert scale, and the last 2 items were responded to as "have not had symptoms," 0 (I did not recognize the symptoms), 1 (not quickly) to 5 (very quickly), and Self-Care Management (5-point Likert scale from 1 to 5 for the first 7 items and a 6-point rating scale for the last item). Symptom perception was found to include monitoring ("listening" to their bodies) and recognition (engage in active behaviors based on interpretation of symptoms) of heart failure symptoms.
  Higher total scores indicate higher heart failure self-care and higher sub-scale scores indicate higher maintenance, management, and perception of heart failure.

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic Avon Hospital, Avon, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yilmaz S, Omurlu IK. Survival after cardiopulmonary arrest in a tertiary care hospital in Turkey. Ann Saudi Med. 2019 Mar-Apr;39(2):92-99. doi: 10.5144/0256-4947.2019.07.03.1400. PMID 30905924
- [Background] Virani SS, Alonso A, Aparicio HJ, Benjamin EJ, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Cheng S, Delling FN, Elkind MSV, Evenson KR, Ferguson JF, Gupta DK, Khan SS, Kissela BM, Knutson KL, Lee CD, Lewis TT, Liu J, Loop MS, Lutsey PL, Ma J, Mackey J, Martin SS, Matchar DB, Mussolino ME, Navaneethan SD, Perak AM, Roth GA, Samad Z, Satou GM, Schroeder EB, Shah SH, Shay CM, Stokes A, VanWagner LB, Wang NY, Tsao CW; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2021 Update: A Report From the American Heart Association. Circulation. 2021 Feb 23;143(8):e254-e743. doi: 10.1161/CIR.0000000000000950. Epub 2021 Jan 27. PMID 33501848
- [Background] Spertus JA, Jones PG. Development and Validation of a Short Version of the Kansas City Cardiomyopathy Questionnaire. Circ Cardiovasc Qual Outcomes. 2015 Sep;8(5):469-76. doi: 10.1161/CIRCOUTCOMES.115.001958. PMID 26307129
- [Background] Schneider MA, Howard KA. Using Technology to Enhance Discharge Teaching and Improve Coping for Patients After Stroke. J Neurosci Nurs. 2017 Jun;49(3):152-156. doi: 10.1097/JNN.0000000000000275. PMID 28346312
- [Background] Riegel B, Jaarsma T, Stromberg A. A middle-range theory of self-care of chronic illness. ANS Adv Nurs Sci. 2012 Jul-Sep;35(3):194-204. doi: 10.1097/ANS.0b013e318261b1ba. PMID 22739426
- [Background] Riegel B, Barbaranelli C, Carlson B, Sethares KA, Daus M, Moser DK, Miller J, Osokpo OH, Lee S, Brown S, Vellone E. Psychometric Testing of the Revised Self-Care of Heart Failure Index. J Cardiovasc Nurs. 2019 Mar/Apr;34(2):183-192. doi: 10.1097/JCN.0000000000000543. PMID 30303894
- [Background] Reeder KM, Ercole PM, Peek GM, Smith CE. Symptom perceptions and self-care behaviors in patients who self-manage heart failure. J Cardiovasc Nurs. 2015 Jan-Feb;30(1):E1-7. doi: 10.1097/JCN.0000000000000117. PMID 24335834
- [Background] Quan H, Sundararajan V, Halfon P, Fong A, Burnand B, Luthi JC, Saunders LD, Beck CA, Feasby TE, Ghali WA. Coding algorithms for defining comorbidities in ICD-9-CM and ICD-10 administrative data. Med Care. 2005 Nov;43(11):1130-9. doi: 10.1097/01.mlr.0000182534.19832.83. PMID 16224307
- [Background] Quan H, Li B, Couris CM, Fushimi K, Graham P, Hider P, Januel JM, Sundararajan V. Updating and validating the Charlson comorbidity index and score for risk adjustment in hospital discharge abstracts using data from 6 countries. Am J Epidemiol. 2011 Mar 15;173(6):676-82. doi: 10.1093/aje/kwq433. Epub 2011 Feb 17. PMID 21330339
- [Background] Park LG, Dracup K, Whooley MA, McCulloch C, Jin C, Moser DK, Clark RA, Pelter MM, Biddle M, Howie Esquivel J. Symptom Diary Use and Improved Survival for Patients With Heart Failure. Circ Heart Fail. 2017 Nov;10(11):e003874. doi: 10.1161/CIRCHEARTFAILURE.117.003874. PMID 29158435
- [Background] Negarandeh R, Aghajanloo A, Seylani K. Barriers to Self-care Among Patients with Heart Failure: A Qualitative Study. J Caring Sci. 2020 Oct 20;10(4):196-204. doi: 10.34172/jcs.2020.026. eCollection 2021 Nov. PMID 34849365
- [Background] Musekamp G, Schuler M, Seekatz B, Bengel J, Faller H, Meng K. Does improvement in self-management skills predict improvement in quality of life and depressive symptoms? A prospective study in patients with heart failure up to one year after self-management education. BMC Cardiovasc Disord. 2017 Feb 15;17(1):51. doi: 10.1186/s12872-017-0486-5. PMID 28196523
- [Background] Latorre-Postigo JM, Ros-Segura L, Navarro-Bravo B, Ricarte-Trives JJ, Serrano-Selva JP, Lopez-Torres-Hidalgo J. Older adults' memory for medical information, effect of number and mode of presentation: An experimental study. Patient Educ Couns. 2017 Jan;100(1):160-166. doi: 10.1016/j.pec.2016.08.001. Epub 2016 Aug 21. PMID 27567498
- [Background] Imam Z, Odish F, Gill I, O'Connor D, Armstrong J, Vanood A, Ibironke O, Hanna A, Ranski A, Halalau A. Older age and comorbidity are independent mortality predictors in a large cohort of 1305 COVID-19 patients in Michigan, United States. J Intern Med. 2020 Oct;288(4):469-476. doi: 10.1111/joim.13119. Epub 2020 Jun 22. PMID 32498135
- [Background] Heo S, Moser DK, Lennie TA, Kim J, Turrise S, Troyan PJ, Kang J, Jones HJ. Self-care strategies and interventions needed in patients with heart failure: from patient perspectives-a qualitative study. Eur J Cardiovasc Nurs. 2021 Aug 20;20(6):540-546. doi: 10.1093/eurjcn/zvaa033. PMID 34008023
- [Background] Hagglund E, Lynga P, Frie F, Ullman B, Persson H, Melin M, Hagerman I. Patient-centred home-based management of heart failure. Findings from a randomised clinical trial evaluating a tablet computer for self-care, quality of life and effects on knowledge. Scand Cardiovasc J. 2015 Aug;49(4):193-9. doi: 10.3109/14017431.2015.1035319. Epub 2015 Jun 4. PMID 25968968
- [Background] Greene SJ, Butler J, Spertus JA, Hellkamp AS, Vaduganathan M, DeVore AD, Albert NM, Duffy CI, Patterson JH, Thomas L, Williams FB, Hernandez AF, Fonarow GC. Comparison of New York Heart Association Class and Patient-Reported Outcomes for Heart Failure With Reduced Ejection Fraction. JAMA Cardiol. 2021 May 1;6(5):522-531. doi: 10.1001/jamacardio.2021.0372. PMID 33760037
- [Background] Green CP, Porter CB, Bresnahan DR, Spertus JA. Development and evaluation of the Kansas City Cardiomyopathy Questionnaire: a new health status measure for heart failure. J Am Coll Cardiol. 2000 Apr;35(5):1245-55. doi: 10.1016/s0735-1097(00)00531-3. PMID 10758967
- [Background] Foraker RE, Rose KM, Chang PP, Suchindran CM, McNeill AM, Rosamond WD. Hospital length of stay for incident heart failure: Atherosclerosis Risk in Communities (ARIC) cohort: 1987-2005. J Healthc Qual. 2014 Jan-Feb;36(1):45-51. doi: 10.1111/j.1945-1474.2012.00211.x. Epub 2012 Dec 3. PMID 23206293
- [Background] Cocks K, Torgerson DJ. Sample size calculations for pilot randomized trials: a confidence interval approach. J Clin Epidemiol. 2013 Feb;66(2):197-201. doi: 10.1016/j.jclinepi.2012.09.002. Epub 2012 Nov 27. PMID 23195919
- [Background] Charlson ME, Carrozzino D, Guidi J, Patierno C. Charlson Comorbidity Index: A Critical Review of Clinimetric Properties. Psychother Psychosom. 2022;91(1):8-35. doi: 10.1159/000521288. Epub 2022 Jan 6. PMID 34991091
- [Background] Austin RC, Schoonhoven L, Clancy M, Richardson A, Kalra PR, May CR. Do chronic heart failure symptoms interact with burden of treatment? Qualitative literature systematic review. BMJ Open. 2021 Jul 30;11(7):e047060. doi: 10.1136/bmjopen-2020-047060. PMID 34330858
- [Background] Auld JP, Mudd JO, Gelow JM, Hiatt SO, Lee CS. Self-care Moderates the Relationship Between Symptoms and Health-Related Quality of Life in Heart Failure. J Cardiovasc Nurs. 2018 May/Jun;33(3):217-224. doi: 10.1097/JCN.0000000000000447. PMID 28930784
- [Background] Arbaje AI, Hughes A, Werner N, Carl K, Hohl D, Jones K, Bowles KH, Chan K, Leff B, Gurses AP. Information management goals and process failures during home visits for middle-aged and older adults receiving skilled home healthcare services after hospital discharge: a multisite, qualitative study. BMJ Qual Saf. 2019 Feb;28(2):111-120. doi: 10.1136/bmjqs-2018-008163. Epub 2018 Jul 17. PMID 30018114